CLINICAL TRIAL: NCT02495155
Title: Initial Assessment of an Internet-based Symptom Management Intervention in Early Stage Breast Cancer
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, N. Lynn Henry, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00095498
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Fatigue; Insomnia; Pain
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fatigue (Active Comparator): Participants who have received treatment for early stage breast cancer and who experience fatigue, rated at least a 4 on a scale of 0-10 during the previous week, per patient report. Participants will complete baseline symptom questionnaires, then complete an internet-based cognitive behavioral therapy program (PROSPECT) for 8 weeks, then repeat questionnaires.
  Interventions: Behavioral: PROSPECT
- Treatment-related Pain (Active Comparator): Participants who have received treatment for early stage breast cancer and who experience pain, rated at least a 4 on a scale of 0-10 during the previous week, per patient report. Participants will complete baseline symptom questionnaires, then complete an internet-based cognitive behavioral therapy program (PROSPECT) for 8 weeks, then repeat questionnaires.
  Interventions: Behavioral: PROSPECT
- Insomnia (Active Comparator): Participants who have received treatment for early stage breast cancer and who experience insomnia, assessed as difficulty sleeping over the last week, yes or no, per patient report. Participants will complete baseline symptom questionnaires, then complete an internet-based cognitive behavioral therapy program (PROSPECT) for 8 weeks, then repeat questionnaires.
  Interventions: Behavioral: PROSPECT

INTERVENTIONS:
Behavioral: PROSPECT — PROSPECT is an internet-based exercise and behavioral symptom management program developed for patients who experience long-term side effects from cancer treatment. The cancer-specific symptom management intervention is intended as a self-management adjunct to improve cancer- and treatment-related symptoms through non-pharmacologic approaches.

SUMMARY:
In order to determine the acceptability of a breast cancer-specific cognitive behavioral therapy intervention, as well as to obtain preliminary data to assess efficacy in managing symptoms, the investigators will ask 45 breast cancer survivors with moderate insomnia, fatigue, and/or pain to use the investigators' internet-based intervention for 8 weeks and to complete patient-reported outcomes assessments before and after the 8 week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Stage 0-III invasive carcinoma of the breast
* Surgical resection and axillary assessment, radiation therapy, and/or chemotherapy, as indicated, completed at least 3 months prior to enrollment.
* Concomitant trastuzumab and anti-endocrine therapies are permitted. If taking anti-endocrine therapy must have been taking for at least 3 months prior to enrollment.
* Must report at least one of the following:

  1. Fatigue in the week prior to enrollment at least 4 on a 10 point scale (with 0 = not tired at all and 10 = extremely tired)
  2. Insomnia in the week prior to enrollment
  3. Pain in the week prior to enrollment at least 4 on a 10 point scale (with 0 = no pain and 10 = extremely severe pain)
* Has access to and is able to operate a computer with internet access.
* Able to read and understand English.
* Willing and able to sign an informed consent document.

Exclusion Criteria:

- Diagnosis of sleep apnea or restless leg syndrome that is currently interfering with sleep

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Improvement in patient-reported symptom with use of PROSPECT for 8 weeks | 8 weeks
  To obtain preliminary data about the efficacy of the intervention in this patient population. The investigators will assess change in the participant's primary reported symptom (pain, insomnia, or fatigue) with 8 weeks of the intervention.

SECONDARY OUTCOMES:
Acceptability of the PROSPECT intervention based on patient self-report | 8 weeks
  To obtain preliminary data about the acceptability and usability of the intervention in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- See also: for information about clinical trials at University of Michigan, including this one — http://www.mcancer.org/about/cancer-answerline